CLINICAL TRIAL: NCT05898958
Title: Impact of Ultrasound-Guided Rhomboid Intercostal and Sub-Serratus Block Versus Thoracic Paravertebral Block on Improving Pulmonary Functions for Multiple Rib Fractures
Brief Title: Rhomboid Intercostal and Sub-Serratus Block for Improving Pulmonary Function and Pain in Patients With Fracture Ribs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ahmed Raafat Mansour Saif Elbalat, Assistant lecturer in anesthesia,icu and pain department, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9001-17-10-2021
Record Dates: First submitted 2023-05-14; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Fracture Rib
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- I.v morphine infusion (No Intervention): A loading i.v. dose of 0.15 mg/kg morphine sulphate diluted in 10 ml of normal saline was given slowly over4-5 min. Then, the morphine infusion will be started bysyringe pump in a dose of 0.05 mg/kg/h that wastitrated to keep the VAS less than 3 at rest andRamsay Sedation Scale (RSS) up to 4
- Thoracic paravertebral block(TPVB) (Experimental): Procedure/Surgery: thoracic paravertebral block The block will be performed in the lateral position.After skin sterilization,the ultrasound transducerprobe (6-13-MHz high-frequency linear transducer) is positioned in the vertical plane ∼2.5 cm lateral tomarked spinous process with its orientation directedcranially. T.After local anesthetic infiltration, an 18-gauge Tuohy needle will be inserted into the paravertebral spacein an 'in plane' technique. After a negativeaspiration through the needle, 20 ml of 0.25%bupivacaine with 1: 200 000 epinephrine will be injected slowly over 3 min.A20-G epidural catheter will be threaded through Tuohyneedle and advanced 2-3 cm into the paravertebral space.Anyprocedure-related adverse effects will be noted, and thedermatomal loss of pin prick sensation will be testedover both sides.
  Interventions: Procedure: thoracic paravertebral block
- Rhomboid Intercostal , subserratus block (RISSB) (Experimental): The ultrasound probe will be placed in the obliquesagittal plane orientation, 1-2 cm medial to the medial scapula at theT5-T6 level. The trapezius muscle, rhomboid major muscle, ribs, intercostal muscle and pleura will be visualized respectively using ultrasound.After local anesthetic infiltration, needle will be inserted from the cranial to the caudal direction using the in-plane technique. The needle will be advanced between the rhomboid major and intercostal muscle fascia. The location of the needle will be confirmed with 2 mL saline solution, 10 ml of 0.25% bupivacaine with 1 : 200 000 epinephrine will beinjected slowly over 3min.for the subserratus block 10 ml of 0.25%bupivacaine with 1 : 200 000 epinephrine will be injected betweenthe serratus and intercostal muscle fascia at level of t9.
  Interventions: Procedure: rhomboid intercostal and subserratus block

INTERVENTIONS:
Procedure: thoracic paravertebral block — The block will be performed in the lateral position.After skin sterilization,the ultrasound transducerprobe (6-13-MHz high-frequency linear transducer) is positioned in the vertical plane ∼2.5 cm lateral tomarked spinous process with its orientation directedcranially. T.After local anesthetic infiltration, an 18-gauge Tuohy needle will be inserted into the paravertebral spacein an 'in plane' technique. After a negativeaspiration through the needle, 20 ml of 0.25%bupivacaine with 1: 200 000 epinephrine will be injected slowly over 3 min.A20-G epidural catheter will be threaded through Tuohyneedle and advanced 2-3 cm into the paravertebral space.Anyprocedure-related adverse effects will be noted, and thedermatomal loss of pin prick sensation will be testedover both sides.
  Arms: Thoracic paravertebral block(TPVB)
Procedure: rhomboid intercostal and subserratus block — The ultrasound probe will be placed in the obliquesagittal plane orientation, 1-2 cm medial to the medial scapula at theT5-T6 level. The trapezius muscle, rhomboid major muscle, ribs, intercostal muscle and pleura will be visualized respectively using ultrasound.After local anesthetic infiltration, needle will be inserted from the cranial to the caudal direction using the in-plane technique. The needle will be advanced between the rhomboid major and intercostal muscle fascia. The location of the needle will be confirmed with 2 mL saline solution, 10 ml of 0.25% bupivacaine with 1 : 200 000 epinephrine will beinjected slowly over 3min.for the subserratus block 10 ml of 0.25%bupivacaine with 1 : 200 000 epinephrine will be injected betweenthe serratus and intercostal muscle fascia at level of t9.
  Arms: Rhomboid Intercostal , subserratus block (RISSB)

SUMMARY:
Rib fractures are seen in more than 50% of patient spresenting with blunt chest trauma and are associated with significant morbidity, long-term disability and mortality .

Many of these adverse consequences are a result ofinadequately controlled pain which hinders respiration,leading to atelectasis, pneumonia and respiratory failure .

The early provision of adequate analgesia is thereforeparamount in the management of these patients. The cornerstones of analgesic management are oral andintravenous medications such as paracetamol, nonsteroidal anti-inflammatorydrugs(NSAIDs) and opioids.

Nevertheless, in patients with more significant injuries orcomorbidities, interventional procedures are often neededto provide adequate analgesia and avoid opioid-relatedadverse effects .

DETAILED DESCRIPTION:
Paravertebral block (PVB), through injecting a local anaesthetic agent close towhere the spinal nerves exit the intervertebral foramina, can provide high quality ipsilateral, segmental, somatic, and sympathetic nerve blockad.

PVB is a successful regional method for amelioration of pain in patients undergoingesophagectomy, breastsurgery, thoracotomy, cardiacsurgery,hepatectomy,percutaneusnephrolithotomyand nephrectomy .Thoracic paravertebralblock(TPVB) has also been used for pain reliefof multiplerib fractures ( MRFs).

Rhomboid intercostal and sub-serratus block (RISS) is an alternative block for multiple rib fractures.

The rhomboid intercostal block was first described in 2016 . The region described is known as the triangle of auscultation that is bounded medially by inferior part of the trapezius, inferiorly by the superior border oflatissimusdorsi, and laterally by the medial border of the scapula. In this ultrasound-guided block, the local anesthetic drug is administered between the rhomboid major and the intercostal muscle fascia at the level of T6-T7 and provides analgesia of T3-T8 dermatomes .

Elsharkawy et al. described a modification to the rhomboid intercostal block to expand dermatomal coverage fromT2-T11 dermatomes. They describe theRISS (Rhomboid Intercostal and Sub-Serratus) block that is a twoinjection block of both the rhomboidintercostal and sub-serratusspace. After the first injection, theultrasound probe advances caudally and laterally distal to the inferior angle of the scapula, the second injection apply between the serratus and intercostal muscle fascia.

Because comparison betweenTPVB and RISS in patients with MRF has rarely been reported.Therefore, this study aimed to assess theeffect ofRISS on pain managementand pulmonary functions compared with TPVB in patients withMRFs.

ELIGIBILITY:
Inclusion Criteria:

* writteninformedconsentfrom the patient.
* Patient with unilateral multiple rib fractures(≥3fractures). ASA I and II . Age 18-60 years old. Both gender. BMI 25- 30 Kg/m2. Cooperative patients.

Exclusion Criteria:

* Compromised airway. Any trauma in the patient that interfere with the positioning of patients for block.

Patients who needed mechanical ventilation before or during the study. Patients with associated head trauma. Patient with hemodynamic instability and need inotropic support. Patient with abbreviated injury scale (AIS) in extremity more than 2 Peripheral neuropathy. Pathological coagulopathy. Infection at the injection site. Untreated pneumothorax. Disturbed conscious level. An allergy to local anesthetics used in this study. Endocrinaldiseases including DM

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function test FEV1 by using Hand-held spirometry | 3 days
  Spirometry is the most frequently used measure of lung function and is a measure of volume against time . The spirometer will be used to measure pulmonary function tests namely; FEV1 .Forced expiratory volume (FEV1) measure show how much air a person can exhale in a forced breath during the first second.
The visual analog scale (VAS) | 3 days
  The visual analog scale (VAS) will be used to assess pain severity and control. VAS is a simple assessment tool consisting of a 10-cmline, where 0=no pain at all, 1-2=mild pain intensity,3-5=moderate pain intensity, 6-8=severe pain intensity, and 9-10=worst pain was felt.(22)

CONTACTS AND LOCATIONS:
Overall Officials: Sanaa A Eltohamy, Study Director — Zagazig University
Locations (1):
- Zagazig, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No